CLINICAL TRIAL: NCT04691089
Title: Professional Rescuers Cardiopulmonary Resuscitation Performance After Implementation of a Defibrillation Algorithm for Early Treatment of Refibrillation, an Observational Study.
Brief Title: Cardiopulmonary Resuscitation Performance of Professional Rescuers With a New Defibrillation Algorithm
Acronym: DEFI-2022
Status: Completed | Type: Observational
Sponsor: French Defence Health Service (Other Government)
Responsible Party: Principal Investigator, Daniel Jost, Principal Investigator, Fire Brigade Of Paris Emergency Medicine Dept
Other Study IDs: DEFI 2022 OBSERVATIONAL
Record Dates: First submitted 2020-10-31; First posted 2020-12-31 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Arrest, Sudden; Ventricular Tachycardia; Ventricular Fibrillation; Sudden Cardiac Death
Keywords: Cardiac Arrest; Automatic External Defibrillator; Chest Compression Fraction; Electrical Cardiac Analysis under Chest Compressions
MeSH Terms: conditions — Death, Sudden, Cardiac; Tachycardia, Ventricular; Ventricular Fibrillation; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the Paris (France) Medical Emergency system, in the early phase of Out-of-hospital Cardiac Arrest (OHCA), the treatment of a Ventricular Fibrillation (VF) consists of delivering an External Electric Shock (EES) by a rescuer with the use of an Automated External Defibrillator (AED). This latter realizes a cardiac rhythm analysis every two minutes. This analysis requires that chest compressions (CC) be interrupted for a while. However, CC interruptions are potentially harmful due to the brain, and heart perfusions decrease.

On the other hand, the recurrence of VF occurs mostly during the first minute after the shock, whereas the delay between 2 rhythm analysis is 2 minutes. The consequence is excessive time spent in VF, which is deleterious in terms of coronary and cerebral perfusion.

The investigator implements a new AED algorithm whose operating principle is as follows. One minute after an EES administration, the AED realizes a cardiac rhythm analysis during which the rescuers do not need to interrupt the chest compressions (CC): this is called the rhythm analysis " in presence of CC" The detection of a VF " in presence of CC " needs to be confirmed, " in absence of CC " The CC's are therefore interrupted for new rhythm analysis. Once the presence of VF is approved, the AED proposes a shock to be administred

The aim of the study

Study Design:

This is a prospective observational study.

The eligibility criteria are as follows:

* Patients in Out-Of-Hospital Cardiac Arrest.
* Basic Life support care with an AED.

The primary endpoint is the " chest-compression fraction (CCF) " that represents the CPR-time performance during the ten first minutes of BLS care ( or < 10 min in case of Return Of Spontaneus Circulation (ROSC))

DETAILED DESCRIPTION:
BACKGROUND

For Out-Of-Hospital Cardiac Arrest (OHCA) patients suffering from ventricular fibrillation (VF) or ventricular tachycardia (VT), BLS care consists of administering external electric shocks (EES) and cardiopulmonary resuscitation (CPR). However, despite successful defibrillation, VF recurs in 50% of cases. Rescuers are forced to repeat EES as often as needed, without the recommendations specifying a maximum number.

International guidelines recommend a 2-min CPR time between 2 rhythm analysis, that means one shock every 2 min. Since refibrillation occurs mostly during the first-minute post-shock, the patient will have to wait until the end of the 2 minutes before receiving the next EES. During that time, the chest compressions (CC) provide a reduced fraction of physiologic blood flow.

The new AED algorithm provides the following changes :

* After a 60-second post-shock CPR-period, the AED performs an analysis "in presence of CC" i.e., without CC interruption is performed.
* Each time the AED detects a VF "in presence of CC" the algorithm requires the CC to be interrupted to perform an analysis "in absence of CC " to confirm the rhythm shockability.
* Analyses "in presence of CC" are triggered every minute, possibly followed or not by an analysis " in absence of CC "
* at least, the algorithm performs an analysis " in absence of CC " systematically every 2 minutes.

This new algorithm fits in between two historical CPR algorithms used in western medical systems - the one-minute and the two-minute CPR cycle- depending on the rhythm shockability detected " in presence of CC "

OBJECTIVES

The main objective is to measure the " CC fraction " during the ten first minutes of Fire Fighter BLS care in OHCA.

The secondary objectives :

1. Report on the available CPR quality parameters (CC frequency, hands-off maximum).
2. Report on the AED's diagnostic performance when analyzing the rhythm "in presence of CC "
3. Report on the AED's diagnostic performance when analyzing the rhythm " in absence of CC "
4. Report on the overall AED's diagnostic performance that results from the combination of two consecutive analyses " in presence of CC " and " in absence of CC"
5. Report on post-shock rhythms and their incidence
6. Report on the number of EES per patient
7. Report on the time distribution for the shocks administered per-patient to describe the rhythmic storm.
8. Report on the incidence of Return Of Spontaneous Circulation (ROSC), survival at hospital admission, and survival at hospital discharge.
9. Compare these reports to a historical cohort (2017).

METHOD

This is a prospective observational study.

* The observation window is limited to CPR cycles within the first 10 minutes of BLS care, or less if ROSC is presumed.
* The choice of 10 minutes is intended to observe the BLS team's action, without interfering with the ALS team that arrives later.
* The three following criteria define a presumptive ROSC:
* 1. presence of QRS complexes of broadly similar morphology
* 2. synchronous impedance curve variation with the QRS complexes (indicating intrathoracic movement, in that case, cardiac mechanical activity)
* 3. no on-going CC
* A CPR cycle is defined by the delay between two " in absence of CC " analyses.

The study does not imply any change in current practice. There is no planned interim analysis.

All consecutive participants with inclusion criteria and no exclusion criteria will be analyzed.

STUDY SIZE

The sample size was calculated to perform a non-inferiority analysis first, followed by a superiority test if non-inferiority was demonstrated.

Non-inferiority test. The formula for calculating the required sample size in each group is based on a well-established statistical methodology designed for comparing two means in the context of a non-inferiority test.

n = ((Z α/2 + Z β)2 X (σ12 + σ22)) / (μ1- μ2 - δ)2

With:

* Sample size (n): the number of subjects required in each group.
* α risk: Initially set at 0.025, this value is adjusted to account for multiple hypothesis testing by applying the Bonferroni correction.
* Power 1- β: Established at 90%
* Expected mean difference: This value is set to zero for this study.
* σ (Standard Deviation): The value for each group has been set to 17.
* δ (Non-Inferiority Margin): This margin is set at 5, an arbitrary value considered the maximal loss of effect (inferiority) that would be clinically acceptable when comparing CCF 2021 with CCF 2017

After the calculations, the required sample size was 208 subjects for each group involved in the non-inferiority testing.

Superiority test. Should the non-inferiority hypothesis not be rejected, the study design allows for a subsequent superiority test to be conducted.

For superiority, the investigators use the formula :

n = ((Z α/2 + Z β)2 X (σ12 + σ22)) / (μ1- μ2)2

With:

* Z α/2 : the Z value for an alpha/2 significance level
* Z β : the Z value for a 1-beta power
* σ12 and σ22 : the variances of the two groups
* μ1 and μ2 : the means of the two groups.

For α risk = 0.025 (Bonferroni correction), a power established at 90%, a standard deviation of 17, and a detectable difference between the two groups of 5%, the required sample size was 256 subjects for each group involved in the superiority testing. (STATA : sampsi 65 70 ,SD(17) alpha(0.025)) To account for a 10% loss of subjects, the number of patients was increased to 282, rounded up to 285 per group, i.e., a total of 570 patients.

To observe 285 shockable patients, the investigators estimate the observation time required to be one year.

Note that this same number of patients will be sufficient to detect an absolute 10% difference with an alpha risk of 5% and a power of 90%, between patients in the "2017" group and patients in the "2020" group with regard to the secondary endpoint "Survival at hospital admission"

INTERRUPTION OR STOPPING OF THE STUDY

The sponsor has the responsibility to report, to the national health authority, any serious and unexpected adverse events attributable to the new AED algorithm.

RISKS

A full report on the risks, the description of incidents, accidents and adverse events will be the subject of a chapter in the results section and also in the discussion.

FINANCING

Funding for the study is provided by the Paris Fire Brigade (promoter, following acceptance of the survey under French policy for clinical research projects)

DISCUSSION

The study will report on the CC fraction of an AED algorithm designed to analyze "under CC."

ELIGIBILITY:
Inclusion Criteria:

-Non-traumatic OHCA in adults, treated by a BLS team and connected to an AED equipped either with the 2017 or with the 2020 algorithm.

Exclusion Criteria:

* Use of AED in a pediatric mode
* CPR administered in 15:2 mode
* Patient already connected to another defibrillator at the arrival of the BLS Team
* No shock advised by defibrillator at first analysis
* Patient with a pacemaker

Secondary Exclusion Criteria

* Surviving patients' opposition to the use of their data.
* Patients with unreadable electrocardiographic or impedance data.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical OHCA patients of the greater Paris (Paris, Haut-de-Seine, Seine-Saint-Denis and Val- de-Marne Country)
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-04-02 (Actual)

PRIMARY OUTCOMES:
Report on Chest Compression Fraction (CCf) | 10 minutes
  CCf is the length of time the patient receives chest compression/management time (describe as a %)

SECONDARY OUTCOMES:
Report on Cardiopulmonary Resuscitation (CPR) parameters : CPR ratio | 10 minutes
  CPR ratio (time during which the patient receives chest compression and bag ventilation / total management time; describe as a %)
Report on Cardiopulmonary Resuscitation (CPR) parameters :Prompt CPR fraction | 10 minutes
  Prompt CPR fraction (duration between the two AED announcements "resume massage" and "interrupt massage"/ total management time; describe as a %)
Report on Cardiopulmonary Resuscitation (CPR) parameters:Maximal Hands-Off time | 10 minutes
  Maximal Hands-Off time (longest time frame without any CC; describe in seconds)
Report on Cardiopulmonary Resuscitation (CPR) parameters:Chest Compression Frequency | 10 minutes
  Chest Compression Frequency (i.e., measurement of the mobile frequency over 3 to 5 compressions; describe as number of chest compressions by minute)
Report on the diagnostic performance of the AED algorithms "during CC" and " in absence of CC" | 10 minutes
  Calculate Sensibility and Specificity
Report on the overall diagnostic performance resulting from the combination of the consecutive analyses " in presence of CC " and " in absence of CC" | 10 minutes
  Calculate Sensibility and Specificity
Report on five-second-post-shock rhythms and their incidence | 10 minutes
  asystole, pulseless electrical activity, ventricular tachycardia, ventricular fibrillation for "in absence of CC" analysis, at 5 seconds
Report on 60-second-post-shock rhythms and their incidence | 10 minutes
  asystole, pulseless electrical activity, ventricular tachycardia, ventricular fibrillation for "in absence of CC" analysis, at 60 seconds
Report on 120 second-post-shock rhythms and their incidence | 10 minutes
  asystole, pulseless electrical activity, ventricular tachycardia, ventricular fibrillation for "in absence of CC" analysis, at 120 seconds
Report on 15-second-post-shock rhythms and their incidence | 10 minutes
  asystole, pulseless electrical activity, ventricular tachycardia, ventricular fibrillation for "in absence of CC" analysis, at 15 seconds
Report on 30-second-post-shock rhythms and their incidence | 10 minutes
  asystole, pulseless electrical activity, ventricular tachycardia, ventricular fibrillation for "in absence of CC" analysis, at 30 seconds
Report on the number of electrical shocks (EES) delivered and the duration of the rhythmic storm | 1 hour
  Total number of EES delivered (describe as a number)
Report on the number of electrical shocks (EES) intended and the duration of the rhythmic storm | 1 hour
  Ratio "number of EES intended / number of EES delivered" (describe as a ratio %)
Report on the temporal distribution of electrical shocks (EES) and the duration of the rhythmic storm | 1 hour
  EES temporal distribution per patient
Report on the delay from start to end of cumulative VF episodes | 1 hour
  The time period from the start of the first occurence of VF to to the ending of the last episode of ventricular fibrillation (VF) ( seconds)
The time period from the AED-switch-on and the first EES (describe in seconds) | 1 hour
  The time period from the AED-switch-on and the first EES (describe in seconds)
The distribution over time of EES. | 1 hour
  The distribution over time of EES.
Outcomes - ROSC | 2 hours
  Return Of Spontaneous Circulation (ROSC) (describe as a ratio of patients with ROSC / patients included)
Outcomes - admitted alive at hospital | 2 hours
  Survival to hospital admission (describe as a ratio of patients admitted beating heart to hospital / patients included)
Outcomes - discharged from hospital | 1 month
  Survival at hospital discharge (describe as a ratio of patients discharged alive from hospital / patients included)
Compare Chest Compression Fraction (CCf) to Paris Fire Brigade 2017 historical data | 10 minutes
  CCf is the length of time the patient receives chest compression/management time (describe as a %)
Prompt CPR fraction (duration between the two AED announcements "resume massage" and "interrupt massage"/ total management time; describe as a %) | 10 minutes
  Prompt CPR fraction (duration between the two AED announcements "resume massage" and "interrupt massage"/ total management time; describe as a %)
CPR ratio (time during which the patient receives chest compression and bag ventilation / total management time; describe as a %) | 10 minutes
  CPR ratio (time during which the patient receives chest compression and bag ventilation / total management time; describe as a %)
Maximal Hands-Off time (longest time frame without any CC; describe in seconds) | 10 minutes
  Maximal Hands-Off time (longest time frame without any CC; describe in seconds)
Chest Compression Frequency (i.e., measurement of the mobile frequency over 3 to 5 compressions; describe as number of chest compressions by minute) | 10 minutes
  Chest Compression Frequency (i.e., measurement of the mobile frequency over 3 to 5 compressions; describe as number of chest compressions by minute)
Compare Sensibility and Specificity of AED algorithm "during CC" and "in absence of CC" to 2017 algorithm Sensibility and Specificity | 10 minutes
  Compare Sensibility and Specificity of AED algorithm "during CC" and "in absence of CC" to 2017 algorithm Sensibility and Specificity
Compare the overall diagnostic performance resulting from the combination of the consecutive analyses " in presence of CC " and " in absence of CC" to Paris Fire Brigade 2017 historical data | 10 minutes
  Compare the overall diagnostic performance resulting from the combination of the consecutive analyses " in presence of CC " and " in absence of CC" to Paris Fire Brigade 2017 algorithm Sensibility and Specificity
Compare post-shock rhythms and their incidence to Paris Fire Brigade 2017 historical data | 10 minutes
  Compare asystole, pulseless electrical activity, ventricular tachycardia, ventricular fibrillation incidence for "in presence of CC" analysis, at 5 seconds to Paris Fire Brigade 2017 differents rhythms incidences.
Compare post-shock rhythms and their incidence to Paris Fire Brigade 2017 historical data | 10 minutes
  Compare asystole, pulseless electrical activity, ventricular tachycardia, ventricular fibrillation incidence for "in absence of CC" analysis, at 60 seconds to Paris Fire Brigade 2017 differents rhythms incidences.
Compare post-shock rhythms and their incidence to Paris Fire Brigade 2017 historical data | 10 minutes
  Compare asystole, pulseless electrical activity, ventricular tachycardia, ventricular fibrillation incidence for "in absence of CC" analysis, at 120 seconds to Paris Fire Brigade 2017 differents rhythms incidences.
Compare post-shock rhythms and their incidence to Paris Fire Brigade 2017 historical data | 10 minutes
  Compare asystole, pulseless electrical activity, ventricular tachycardia, ventricular fibrillation incidence for "in absence of CC" analysis, at 5 seconds to Paris Fire Brigade 2017 differents rhythms incidences.
Compare number of electrical shocks (EES) and the duration of the rhythmic storm to Paris Fire Brigade 2017 historical data | 10 minutes
  Total number of EES delivered (describe as a number) compare to Paris Fire Brigade 2017 historical data
Compare number of electrical shocks (EES) and the duration of the rhythmic storm to Paris Fire Brigade 2017 historical data | 10 minutes
  EES temporal distribution per patient compare to Paris Fire Brigade 2017 historical data
Compare number of electrical shocks (EES) and the duration of the rhythmic storm to Paris Fire Brigade 2017 historical data | 10 minutes
  The time period from the start of the first to the end of the last ventricular fibrillation (VF) episode (describe in seconds) compare to Paris Fire Brigade 2017 historical data
Compare number of electrical shocks (EES) and the duration of the rhythmic storm to Paris Fire Brigade 2017 historical data | 10 minutes
  The time period from the AED-switch-on and the first EES (describe in seconds) compare to Paris Fire Brigade 2017 historical data
Compare number of electrical shocks (EES) and the duration of the rhythmic storm to Paris Fire Brigade 2017 historical data | 10 minutes
  Compare the distribution over time of EES.to Paris Fire Brigade 2017 historical data
Outcomes - ROSC | 1 hour
  Compare return Of Spontaneous Circulation (ROSC) to Paris Fire Brigade 2017 historical data (describe as a ratio of patients with ROSC / patients included)
Outcomes - admitted alive at hospital | 2 hours
  Compare survival to hospital admission to Paris Fire Brigade 2017 historical data (describe as a ratio of patients admitted beating heart to hospital / patients included)
Outcomes - hospital discharge | 1 month
  Compare survival at hospital discharge to Paris Fire Brigade 2017 historical data (describe as a ratio of patients discharged alive from hospital / patients included)

CONTACTS AND LOCATIONS:
Overall Officials: Clément DERKENNE, MD, Principal Investigator — Paris Fire Brigade
Locations (1):
- Paris Fire Brigade, Paris, Non, Merci, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker PW, Conway J, Cotton C, Ashby DT, Smyth J, Woodman RJ, Grantham H; Clinical Investigators. Defibrillation or cardiopulmonary resuscitation first for patients with out-of-hospital cardiac arrests found by paramedics to be in ventricular fibrillation? A randomised control trial. Resuscitation. 2008 Dec;79(3):424-31. doi: 10.1016/j.resuscitation.2008.07.017. Epub 2008 Nov 4. PMID 18986748
- [Background] Berdowski J, ten Haaf M, Tijssen JG, Chapman FW, Koster RW. Time in recurrent ventricular fibrillation and survival after out-of-hospital cardiac arrest. Circulation. 2010 Sep 14;122(11):1101-8. doi: 10.1161/CIRCULATIONAHA.110.958173. Epub 2010 Aug 30. PMID 20805427
- [Background] Berdowski J, Tijssen JG, Koster RW. Chest compressions cause recurrence of ventricular fibrillation after the first successful conversion by defibrillation in out-of-hospital cardiac arrest. Circ Arrhythm Electrophysiol. 2010 Feb;3(1):72-8. doi: 10.1161/CIRCEP.109.902114. Epub 2009 Dec 30. PMID 20042768
- [Background] Bobrow BJ, Clark LL, Ewy GA, Chikani V, Sanders AB, Berg RA, Richman PB, Kern KB. Minimally interrupted cardiac resuscitation by emergency medical services for out-of-hospital cardiac arrest. JAMA. 2008 Mar 12;299(10):1158-65. doi: 10.1001/jama.299.10.1158. PMID 18334691
- [Background] Caffrey SL, Willoughby PJ, Pepe PE, Becker LB. Public use of automated external defibrillators. N Engl J Med. 2002 Oct 17;347(16):1242-7. doi: 10.1056/NEJMoa020932. PMID 12393821
- [Background] Cheskes S, Schmicker RH, Christenson J, Salcido DD, Rea T, Powell J, Edelson DP, Sell R, May S, Menegazzi JJ, Van Ottingham L, Olsufka M, Pennington S, Simonini J, Berg RA, Stiell I, Idris A, Bigham B, Morrison L; Resuscitation Outcomes Consortium (ROC) Investigators. Perishock pause: an independent predictor of survival from out-of-hospital shockable cardiac arrest. Circulation. 2011 Jul 5;124(1):58-66. doi: 10.1161/CIRCULATIONAHA.110.010736. Epub 2011 Jun 20. PMID 21690495
- [Background] Christenson J, Andrusiek D, Everson-Stewart S, Kudenchuk P, Hostler D, Powell J, Callaway CW, Bishop D, Vaillancourt C, Davis D, Aufderheide TP, Idris A, Stouffer JA, Stiell I, Berg R; Resuscitation Outcomes Consortium Investigators. Chest compression fraction determines survival in patients with out-of-hospital ventricular fibrillation. Circulation. 2009 Sep 29;120(13):1241-7. doi: 10.1161/CIRCULATIONAHA.109.852202. Epub 2009 Sep 14. PMID 19752324
- [Background] Fumagalli F, Silver AE, Tan Q, Zaidi N, Ristagno G. Cardiac rhythm analysis during ongoing cardiopulmonary resuscitation using the Analysis During Compressions with Fast Reconfirmation technology. Heart Rhythm. 2018 Feb;15(2):248-255. doi: 10.1016/j.hrthm.2017.09.003. Epub 2017 Sep 14. PMID 28917561
- [Background] Gliner BE, White RD. Electrocardiographic evaluation of defibrillation shocks delivered to out-of-hospital sudden cardiac arrest patients. Resuscitation. 1999 Jul;41(2):133-44. doi: 10.1016/s0300-9572(99)00040-4. PMID 10488935
- [Background] Hasselqvist-Ax I, Riva G, Herlitz J, Rosenqvist M, Hollenberg J, Nordberg P, Ringh M, Jonsson M, Axelsson C, Lindqvist J, Karlsson T, Svensson L. Early cardiopulmonary resuscitation in out-of-hospital cardiac arrest. N Engl J Med. 2015 Jun 11;372(24):2307-15. doi: 10.1056/NEJMoa1405796. PMID 26061835
- [Background] Hu Y, Tang H, Liu C, Jing D, Zhu H, Zhang Y, Yu X, Zhang G, Xu J. The performance of a new shock advisory algorithm to reduce interruptions during CPR. Resuscitation. 2019 Oct;143:1-9. doi: 10.1016/j.resuscitation.2019.07.026. Epub 2019 Aug 1. PMID 31377393
- [Background] Jost D, Degrange H, Verret C, Hersan O, Banville IL, Chapman FW, Lank P, Petit JL, Fuilla C, Migliani R, Carpentier JP; DEFI 2005 Work Group. DEFI 2005: a randomized controlled trial of the effect of automated external defibrillator cardiopulmonary resuscitation protocol on outcome from out-of-hospital cardiac arrest. Circulation. 2010 Apr 13;121(14):1614-22. doi: 10.1161/CIRCULATIONAHA.109.878389. Epub 2010 Mar 29. PMID 20351239
- [Background] Kerber RE, Becker LB, Bourland JD, Cummins RO, Hallstrom AP, Michos MB, Nichol G, Ornato JP, Thies WH, White RD, Zuckerman BD. Automatic external defibrillators for public access defibrillation: recommendations for specifying and reporting arrhythmia analysis algorithm performance, incorporating new waveforms, and enhancing safety. A statement for health professionals from the American Heart Association Task Force on Automatic External Defibrillation, Subcommittee on AED Safety and Efficacy. Circulation. 1997 Mar 18;95(6):1677-82. doi: 10.1161/01.cir.95.6.1677. PMID 9118556
- [Background] Krasteva V, Jekova I, Dotsinsky I, Didon JP. Shock advisory system for heart rhythm analysis during cardiopulmonary resuscitation using a single ECG input of automated external defibrillators. Ann Biomed Eng. 2010 Apr;38(4):1326-36. doi: 10.1007/s10439-009-9885-9. Epub 2010 Jan 13. PMID 20069371
- [Background] Roh YI, Jung WJ, Hwang SO, Kim S, Kim HS, Kim JH, Kim TY, Kang HS, Lee JS, Cha KC. Shorter defibrillation interval promotes successful defibrillation and resuscitation outcomes. Resuscitation. 2019 Oct;143:100-105. doi: 10.1016/j.resuscitation.2019.08.022. Epub 2019 Aug 20. PMID 31442471
- [Background] Vaillancourt C, Everson-Stewart S, Christenson J, Andrusiek D, Powell J, Nichol G, Cheskes S, Aufderheide TP, Berg R, Stiell IG; Resuscitation Outcomes Consortium Investigators. The impact of increased chest compression fraction on return of spontaneous circulation for out-of-hospital cardiac arrest patients not in ventricular fibrillation. Resuscitation. 2011 Dec;82(12):1501-7. doi: 10.1016/j.resuscitation.2011.07.011. Epub 2011 Jul 18. PMID 21763252
- [Result] Affatato R, Li Y, Ristagno G. See through ECG technology during cardiopulmonary resuscitation to analyze rhythm and predict defibrillation outcome. Curr Opin Crit Care. 2016 Jun;22(3):199-205. doi: 10.1097/MCC.0000000000000297. PMID 27031917
- [Result] van Alem AP, Post J, Koster RW. VF recurrence: characteristics and patient outcome in out-of-hospital cardiac arrest. Resuscitation. 2003 Nov;59(2):181-8. doi: 10.1016/s0300-9572(03)00208-9. PMID 14625108
- [Derived] Didon JP, Jekova I, Frattini B, Menetre S, Derkenne C, Ha VHT, Jost D, Krasteva V. Clinical performance of AED shock advisory system with integrated Analyze Whilst Compressing algorithm for analysis of the ECG rhythm during out-of-hospital cardiopulmonary resuscitation: A secondary analysis of the DEFI 2022 study. Resusc Plus. 2024 Aug 5;19:100740. doi: 10.1016/j.resplu.2024.100740. eCollection 2024 Sep. PMID 39185280